CLINICAL TRIAL: NCT02075073
Title: A Randomised, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Three Formulations of Trastuzumab (SB3, EU Sourced Herceptin® and US Sourced Herceptin®) in Healthy Male Subjects
Brief Title: Pharmacokinetic, Safety, Tolerability and Immunogenicity Study of SB3 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SB3-G11-NHV; 2013-004112-21 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SB3 (Experimental): SB3, single dose of 6 mg/kg via intravenous infusion (study drug)
  Interventions: Biological: SB3
- EU sourced Herceptin® (Active Comparator): EU sourced Herceptin®, single dose of 6 mg/kg via intravenous infusion (reference drug)
  Interventions: Biological: EU sourced Herceptin®
- US sourced Herceptin® (Active Comparator): US sourced Herceptin®, single dose of 6 mg/kg via intravenous infusion (reference drug)
  Interventions: Biological: US sourced Herceptin®

INTERVENTIONS:
Biological: SB3
  Arms: SB3
Biological: EU sourced Herceptin®
  Arms: EU sourced Herceptin®
Biological: US sourced Herceptin®
  Arms: US sourced Herceptin®

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety, tolerability and immunogenicity of SB3 and Herceptin® (EU sourced Herceptin® and US sourced Herceptin®) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Have a body weight between 60.0 and 94.9 kg and a body mass index between 18.0 and 29.9 kg/m², inclusive.

Exclusion Criteria:

* history of and/or current clinically significant gastrointestinal, renal, hepatic, cardiovascular, haematological (including pancytopenia, aplastic anaemia or blood dyscrasia), pulmonary, neurologic, metabolic (including known diabetes mellitus), psychiatric or significant allergic disease excluding mild asymptomatic allergies.
* history of and/or current cardiac disease
* previously received any monoclonal antibody or fusion protein.
* history of cancer including lymphoma, leukaemia and skin cancer.
* Have received live vaccine(s) within 30 days prior to Screening or who will require a vaccine(s) between Screening and the End of Study visit.
* intake medication with a half-life > 24 h within 1 month or 10 half-lives of the medication prior to the administration of investigational product.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saumsung Bioepis, Study Director — Samsung Bioepis Co., Ltd.
Locations (1):
- Samsung Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Pivot X, Curtit E, Lee YJ, Golor G, Gauliard A, Shin D, Kim Y, Kim H, Fuhr R. A Randomized Phase I Pharmacokinetic Study Comparing Biosimilar Candidate SB3 and Trastuzumab in Healthy Male Subjects. Clin Ther. 2016 Jul;38(7):1665-1673.e3. doi: 10.1016/j.clinthera.2016.06.002. Epub 2016 Jun 29. PMID 27368117

RESULTS

PARTICIPANT FLOW:
Groups:
- SB3 (Proposed Trastuzumab Biosimilar): SB3, single dose of 6 mg/kg via intravenous infusion (study drug)
  SB3
- EU Sourced Herceptin®: EU sourced Herceptin®, single dose of 6 mg/kg via intravenous infusion (reference drug)
  EU sourced Herceptin®
- US Sourced Herceptin®: US sourced Herceptin®, single dose of 6 mg/kg via intravenous infusion (reference drug)
  US sourced Herceptin®
Period: Overall Study
Arm/Group | SB3 (Proposed Trastuzumab Biosimilar) | EU Sourced Herceptin® | US Sourced Herceptin®
Started | 36 | 37 | 36
Completed | 36 | 36 | 36
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB3 (Proposed Trastuzumab Biosimilar) | EU Sourced Herceptin® | US Sourced Herceptin® | Total
Number analyzed (Participants) | 36 | 37 | 36 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.29) | 39.3 (10.80) | 38.7 (11.40) | 38.8 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 36 | 37 | 36 | 109

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Time Frame: 57 days
Measure: Mean (Standard Deviation); unit: µg·h/mL
Arm/Group | SB3 (Proposed Trastuzumab Biosimilar) | EU Sourced Herceptin® | US Sourced Herceptin®
Number analyzed (Participants) | 36 | 36 | 36
µg·h/mL | 34783.4 (5614.13) | 35889.9 (5761.37) | 37370.3 (5620.05)

2. Primary Outcome: Maximum Serum Concentration (Cmax)
Time Frame: 57 days
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | SB3 (Proposed Trastuzumab Biosimilar) | EU Sourced Herceptin® | US Sourced Herceptin®
Number analyzed (Participants) | 36 | 36 | 36
µg/mL | 154.224 (28.0068) | 153.479 (24.7249) | 155.513 (25.5812)

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Time Frame: 57 days
Measure: Mean (Standard Deviation); unit: µg·h/mL
Arm/Group | SB3 (Proposed Trastuzumab Biosimilar) | EU Sourced Herceptin® | US Sourced Herceptin®
Number analyzed (Participants) | 36 | 36 | 36
µg·h/mL | 34320.8 (5349.12) | 35367.5 (5524.09) | 36690.4 (5341.68)

4. Secondary Outcome: Time to Cmax (Tmax)
Time Frame: 57 days
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | SB3 (Proposed Trastuzumab Biosimilar) | EU Sourced Herceptin® | US Sourced Herceptin®
Number analyzed (Participants) | 36 | 36 | 36
hour | 4.691 (15.6597) | 3.529 (7.6948) | 2.799 (3.7569)

ADVERSE EVENTS:
Arm/Group | SB3 (Proposed Trastuzumab Biosimilar) | EU Sourced Herceptin® | US Sourced Herceptin®
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 25/36 | 23/36 | 25/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB3 (Proposed Trastuzumab Biosimilar) (N=36) | EU Sourced Herceptin® (N=36) | US Sourced Herceptin® (N=36)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB3 (Proposed Trastuzumab Biosimilar) (N=36) | EU Sourced Herceptin® (N=36) | US Sourced Herceptin® (N=36)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 1 (1) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (3) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (9) | 8 (8) | 16 (16)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (12) | 4 (4) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Project results may not be published or referred to, in whole or in part, by the Service Provider or any of its Affiliates without the prior expressed written consent of Sponsor, which will not be unreasonably withheld or delayed. Neither Party shall use the other Party's name in connection with any publication or promotion without the other Party's prior written consent.